CLINICAL TRIAL: NCT02524145
Title: Determinants of Chronotropic Incompetence in Patients With Heart Failure and a Preserved Ejection Fraction (HFpEF)
Brief Title: Chronotropic Incompetence in Patients With HFpEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin Levine, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STU 092012-010
Record Dates: First submitted 2015-08-10; First posted 2015-08-14 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Dexmedetomidine; Glycopyrrolate; Isoproterenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Healthy Seniors (Active Comparator): Fifteen healthy senior volunteers > 60 years of age. Subjects will be healthy with no chronic medical problems and on no cardiac medications except for statins. All control subjects will have a Body Mass Index (BMI) <30, with exercise histories of less than 3 days per week of aerobic exercise.
  Intervention: Static handgrip and Autonomic Blockade (Dexmedetomidine, Glycopyrrolate, Isoproterenol)
  Interventions: Other: Static Handgrip; Drug: Dexmedetomidine; Drug: Glycopyrrolate; Drug: Isoproterenol
- HFpEF (Experimental): Patients with HFpEF will provide data from their cardiologist or primary care physician that confirm the following: a) signs and symptoms of heart failure; b) an ejection fraction > 0.50; and c) objective evidence of diastolic dysfunction.
  Intervention: Static handgrip and Autonomic Blockade (Dexmedetomidine, Glycopyrrolate, Isoproterenol)
  Interventions: Other: Static Handgrip; Drug: Dexmedetomidine; Drug: Glycopyrrolate; Drug: Isoproterenol
- Healthy Young (Active Comparator): Fifteen volunteers <45 yrs will be enrolled. Subjects will be healthy with no chronic medical problems and on no cardiac medications except for statins and have BMI <30.
  Intervention: Autonomic Blockade (Dexmedetomidine, Glycopyrrolate, Isoproterenol)
  Interventions: Drug: Dexmedetomidine; Drug: Glycopyrrolate; Drug: Isoproterenol

INTERVENTIONS:
Other: Static Handgrip — Subjects will perform static handgrip at 40% of maximum voluntary contraction until fatigue.
  Arms: HFpEF; Healthy Seniors
Drug: Dexmedetomidine — Subjects will be given dexmedetomidine to suppress sympathetic outflow to minimize sympathetic control over resting heart rate. Subjects will then be given glycopyrrolate to suppress parasympathetic tone to minimize parasympathetic control over resting heart rate. After achievement of autonomic blockade, cardiac beta receptor sensitivity will be assessed by graded infusions of isoproterenol until heart rate increases 30 beats above baseline.
  Other Names: Sympathetic blockade
Drug: Glycopyrrolate — Subjects will be given dexmedetomidine to suppress sympathetic outflow to minimize sympathetic control over resting heart rate. Subjects will then be given glycopyrrolate to suppress parasympathetic tone to minimize parasympathetic control over resting heart rate. After achievement of autonomic blockade, cardiac beta receptor sensitivity will be assessed by graded infusions of isoproterenol until heart rate increases 30 beats above baseline.
  Other Names: Parasympathetic blockade
Drug: Isoproterenol — Subjects will be given dexmedetomidine to suppress sympathetic outflow to minimize sympathetic control over resting heart rate. Subjects will then be given glycopyrrolate to suppress parasympathetic tone to minimize parasympathetic control over resting heart rate. After achievement of autonomic blockade, cardiac beta receptor sensitivity will be assessed by graded infusions of isoproterenol until heart rate increases 30 beats above baseline.
  Other Names: Beta-receptor sensitivity testing

SUMMARY:
The purpose of this study is to determine the mechanisms of chronotropic incompetence (inability to increase heart rate with exercise) in patients with heart failure and preserved ejection fraction (HFpEF). The investigators will test both central command regulation and cardiac beta-receptor sensitivity over control of heart rate.

DETAILED DESCRIPTION:
About half of all elderly patients with a diagnosis of congestive heart failure have apparently normal systolic function, so called "heart failure with a preserved ejection fraction" or HFpEF. To date, no effective therapy for HFpEF has been found, in part because of failure to discern key pathophysiologic pathways.

Although HFpEF is a complex disease with multiple pathophysiologic pathways leading to the phenotype of heart failure, virtually all proposed mechanisms involve some impairment of diastolic function - the inability of the heart to fill adequately at a low enough pressure to avoid congestion which during physical activity or exercise, prevent an increase in heart rate. A number of studies have purported the inability to increase heart rate (chronotropic incompetence) is responsible for the diminished exercise capacity.

Alternatively, the investigators hypothesize that the stiff, slowly relaxing heart of patients with HFpEF causes a marked elevation in pulmonary capillary pressure during exercise which leads to premature fatigue prior to achieving maximal heart rate, thus causing apparent "chronotropic incompetence".

ELIGIBILITY:
Healthy Controls

Inclusion Criteria:

* ages > 60 years
* body mass index <30
* absence of co-morbid conditions including hypertension, diabetes, heart failure, asthma, chronic obstructive pulmonary disease, coronary artery disease as evidenced by angina or prior myocardial infarction or cerebrovascular disease as evidenced by prior transient ischemic attack or stroke

Exclusion Criteria:

* ages less than 60
* body mass index >30
* presence of co-morbid conditions including hypertension, diabetes, heart failure, asthma, chronic obstructive pulmonary disease, coronary artery disease as evidenced by angina or prior myocardial infarction or cerebrovascular disease as evidenced by prior transient ischemic attack or stroke
* Patients with chronic orthopedic injury that might make them unable to participate in an exercise testing will also be excluded
* Subjects unable to speak English will not be recruited because of the complex experimental studies and the need for precise communication between the volunteers and the research staff to ensure safety.

HFpEF Subjects

Inclusion Criteria:

* Patients will be > 60 years old, male or female, all races.
* signs and symptoms of heart failure
* ejection fraction > 0.50
* objective evidence of diastolic dysfunction.
* All patients must be in sinus rhythm without a left bundle branch block at the time of study

Exclusion Criteria:

* underlying valvular or congenital heart disease
* restrictive or infiltrative cardiomyopathy
* acute myocarditis
* New York Heart Association (NYHA) Class IV congestive heart failure, or heart failure that cannot be stabilized on medical therapy
* other condition that would limit the patient's ability to complete the protocol
* manifest ischemic heart disease
* Coumadin/warfarin therapy
* Patients with chronic orthopedic injury that might make them unable to participate in an exercise testing will also be excluded
* Subjects unable to speak English will not be recruited because of the complex experimental studies and the need for precise communication between the volunteers and the research staff to ensure safety.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Levine, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

REFERENCES:
- [Derived] Sarma S, Stoller D, Hendrix J, Howden E, Lawley J, Livingston S, Adams-Huet B, Holmes C, Goldstein DS, Levine BD. Mechanisms of Chronotropic Incompetence in Heart Failure With Preserved Ejection Fraction. Circ Heart Fail. 2020 Mar;13(3):e006331. doi: 10.1161/CIRCHEARTFAILURE.119.006331. Epub 2020 Mar 13. PMID 32164435

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment initiated in June 2015 and completed October 2017. Subjects were recruited from academic medical center cardiology clinic. Healthy control subjects were recruited from the community.
Groups:
- Healthy Seniors: Fifteen healthy senior volunteers > 60 years of age. Subjects will be healthy with no chronic medical problems and on no cardiac medications except for statins.
  Intervention: Static handgrip and Autonomic Blockade (Dexmedetomidine, Glycopyrrolate, Isoproterenol)
  Static Handgrip: Subjects will perform static handgrip at 40% of maximum voluntary contraction until fatigue.
  Autonomic Blockade: Subjects will be given dexmedetomidine and glycopyrrolate to suppress neural control over heart rate during isoproterenol infusion.
- HFpEF: Patients with HFpEF will provide data from their cardiologist or primary care physician that confirm the following: a) signs and symptoms of heart failure; b) an ejection fraction > 0.50; and c) objective evidence of diastolic dysfunction.
  Intervention: Static handgrip and Autonomic Blockade (Dexmedetomidine, Glycopyrrolate, Isoproterenol)
  Static Handgrip: Subjects will perform static handgrip at 40% of maximum voluntary contraction until fatigue.
  Autonomic Blockade: Subjects will be given dexmedetomidine and glycopyrrolate to suppress neural control over heart rate during isoproterenol infusion.
- Healthy Young: Fifteen volunteers <45 yrs will be enrolled. Subjects will be healthy with no chronic medical problems and on no cardiac medications except for statins and have BMI <30.
  Intervention: Autonomic Blockade (Dexmedetomidine, Glycopyrrolate, Isoproterenol)
  Autonomic Blockade: Subjects will be given dexmedetomidine and glycopyrrolate to suppress neural control over heart rate during isoproterenol infusion.
Period: Overall Study
Arm/Group | Healthy Seniors | HFpEF | Healthy Young
Started | 15 | 15 | 10
Completed | 13 | 13 | 7
Not Completed | 2 | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Seniors | HFpEF | Healthy Young | Total
Number analyzed (Participants) | 15 | 15 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 6 | 10 | 17
  >=65 years | 14 | 9 | 0 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Two senior controls, three young controls and two HFpEF subjects withdrew consent.
  years
    number analyzed (Participants) | 13 | 13 | 7 | 33
    (all) | 71 (4) | 68 (6) | 31 (4) | 61 (17)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Two senior controls, three young controls and two HFpEF subjects withdrew consent.
  Participants
    number analyzed (Participants) | 13 | 13 | 7 | 33
    Female | 6 | 7 | 1 | 14
    Male | 7 | 6 | 6 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two senior controls, three young controls and two HFpEF subjects withdrew consent.
  Participants
    number analyzed (Participants) | 13 | 13 | 7 | 33
    Hispanic or Latino | 0 | 1 | 1 | 2
    Not Hispanic or Latino | 13 | 12 | 6 | 31
    Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Two senior controls, three young controls and two HFpEF subjects withdrew consent.
  Participants
    number analyzed (Participants) | 13 | 13 | 7 | 33
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 1 | 2 | 1 | 4
    White | 12 | 11 | 4 | 27
    More than one race | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 10 | 40
Exercise heart rate [Mean (Standard Deviation); unit: beats per minute] — Population: Two senior control, three young control and two HFPEF subjects withdrew after consent.
  beats per minute
    number analyzed (Participants) | 13 | 13 | 7 | 33
    (all) | 156 (15) | 117 (15) | 190 (8) | 148 (32)
Beta-receptor function [Mean (Standard Deviation); unit: beats per ng/kg/min] — Population: Two senior controls, three young controls and two HFpEF subjects withdrew consent
  beats per ng/kg/min
    number analyzed (Participants) | 13 | 13 | 7 | 33
    (all) | 0.254 (0.166) | 0.156 (0.133) | 0.365 (0.129) | 0.239 (0.163)

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Beta-receptor Sensitivity
Description: Cardiac beta-receptor sensitivity will be measured by calculating slope of heart rate versus isoproterenol serum level.
Time Frame: 1 day; primary outcome was complete for each subject in 1 day
Measure: Mean (Standard Deviation); unit: beats per ng/kg/min ISO
Groups:
- Healthy Seniors: Fifteen healthy senior volunteers > 60 years of age. Subjects will be healthy with no chronic medical problems and on no cardiac medications except for statins. All control subjects will have a Body Mass Index (BMI) <30, with exercise histories of less than 3 days per week of aerobic exercise.
  Intervention: Static handgrip and Autonomic Blockade (Dexmedetomidine, Glycopyrrolate, Isoproterenol)
  Static Handgrip: Subjects will perform static handgrip at 40% of maximum voluntary contraction until fatigue.
  Autonomic Blockade: Subjects will be given dexmedetomidine and glycopyrrolate to suppress neural control over heart rate during isoproterenol infusion.
Arm/Group | Healthy Seniors | HFpEF | Healthy Young
Number analyzed (Participants) | 13 | 13 | 7
beats per ng/kg/min ISO | 0.254 (0.166) | 0.156 (0.133) | 0.365 (0.129)

2. Primary Outcome: Central Command Regulation of Heart Rate
Description: Heart rate response to static hand grip immediately followed by supra-systolic arm occlusion and release will determine adequacy on central command control over heart rate response during exercise.
Time Frame: 1 day; primary outcome was complete for each subject in 1 day
Population: Young subjects did not perform handgrip portion of the study.
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Healthy Seniors | HFpEF
Number analyzed (Participants) | 15 | 15
beats per minute | 93 (11) | 89 (14)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Healthy Seniors | HFpEF | Healthy Young
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/7
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2014-12-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT02524145/Prot_000.pdf